CLINICAL TRIAL: NCT06306989
Title: Observational Clinical Study of Letermovir for Preventing CMV Infection After Allo-HSCT
Status: Recruiting | Type: Observational
Sponsor: Cao Weijie (Other)
Responsible Party: Sponsor-Investigator, Cao Weijie, Associate Professor, Zhengzhou University
Organization: Zhengzhou University (Other)
Other Study IDs: Zhengzhou University
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Letemovir for the Prevention of CMV Infection After Allo-HSCT
MeSH Terms: interventions — letermovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-risk groups
  Interventions: Drug: Letermovir
- Low to medium risk group
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Participants will be categorized into high-risk and intermediate-risk groups based on risk factors for CMV infection.Initiate letemovir prophylaxis on day +1 in high-risk patients and on days +7 to +14 in non-high-risk patients.(240 mg, qd in patients with concomitant cyclosporine; 480 mg, qd in patients with concomitant tacrolimus) to +100 days. For patients with comorbid GVHD who require intensive immunosuppression, consider extending the regimen to +200 days.

SUMMARY:
The goal of this observational study is to get a series of clinical data related to the prevention of CMV infection after allo-HSCT with letemovir. The main question it aims to answer are:

* Efficacy and safety of letemovir for the prevention of CMV infection after allo-HSCT.
* Optimal initiation of letemovir to prevent CMV infection. Participants will be categorized into high-risk and intermediate-risk groups based on risk factors for CMV infection.Initiate letemovir prophylaxis on day +1 in high-risk patients and on days +7 to +14 in non-high-risk patients.(240 mg, qd in patients with concomitant cyclosporine; 480 mg, qd in patients with concomitant tacrolimus) to +100 days. For patients with comorbid GVHD who require intensive immunosuppression, consider extending the regimen to +200 days.Treatments they will be given and use bullets.

DETAILED DESCRIPTION:
This observational study was conducted by collecting patients who underwent hematopoietic stem cell transplantation in the Department of Hematology of the First Affiliated Hospital of Zhengzhou University from September 2023 and had IgG-positive CMV serological status, according to whether they had combined risk factors for CMV infection: haploidentical transplantation; umbilical cord blood transplantation; pretreatment regimen of PT-Cy or regimen containing ATG; unrelated donor transplantation; and donor-recipient serological status of D-/R+; Age greater than or equal to 40 years; application of high-dose glucocorticoids (prednisone ≥ 1 mg/kg.d-1 for ≥ 5 days); comorbidities of degree II or greater aGVHD; and division into high-risk and standard-risk groups with different letermovir initiation regimens: letermovir prophylaxis was initiated on day +1 in high-risk patients and on days +7 to +14 in non-high-risk patients (patients with concomitant cyclosporine application, 240 mg. (240 mg, qd, for patients with concomitant cyclosporine; 480 mg, qd, for patients with concomitant tacrolimus) to +100 days, in order to compare the therapeutic benefits of a letemovir-initiated prophylaxis regimen in patients with different risks of infection. After transplantation, blood specimen RT-qPCR was applied once or twice a week for CMV viremia testing, which lasted until 100 days post-transplantation, and it was recommended to appropriately prolong the length of monitoring and shorten the testing interval for high-risk groups.CMV-DNA positivity, the combination of factors related to rejection, recurrence, and CMV, the dosage of immunosuppressant was adjusted, and the initiation of antiviral therapy (ganciclovir, phosphonoinositide, adenosine, etc.) was initiated, until two consecutive CMV-DNA positive days. until CMV-DNA turned negative twice consecutively; if the CMV-DNA copy number increased two weeks after initiating antiviral therapy, CMV drug resistance gene testing was performed. The data were processed statistically using SPSS 25.0 software, the chi-square test was used for categorical measures, and the Nsnn-Whitrey U test was used for continuous variables.OS, EFS, and PFS were analyzed by the log-rank test using the Kaplan-Meier method and survival curves were plotted.Primary study endpoints: incidence of +100-day CMVemia, CMV disease; secondary study endpoints:(1) +30-day CMVemia, CMV disease; +30-day overall survival, non-relapse mortality; +30-day relapse rate; +30-day aGVHD incidence; (2) +100-day overall survival, non-relapse mortality; +100-day relapse rate; +100-day aGVHD incidence;(3) +180 days CMVemia, CMV disease; +180 days overall survival, non-relapse mortality; +180 days relapse rate; +180 days cGVHD incidence.

ELIGIBILITY:
Inclusion Criteria:

1. Biological age not less than 14 years.
2. Positive CMV serology.
3. No detectable CMV-DNA from plasma samples taken 5 days prior to randomization into groups.

Exclusion Criteria:

1. severe hepatic impairment;
2. estimated creatinine clearance of less than 10 ml/min;
3. current or recent recipients of antiviral medications with anti-CMV activity; and
4. any other factor that affects the impact of obtaining data.

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent hematopoietic stem cell transplantation at the Department of Hematology, the First Affiliated Hospital of Zhengzhou University, Zhengzhou, China
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of CMV viremia and CMV disease within 100 days after allogeneic hematopoietic stem cell transplantation. | within 100 days after allogeneic hematopoietic stem cell transplantation
  Prevalence of CMV viremia and CMV disease within 100 days after allogeneic hematopoietic stem cell transplantation.
  [CMV viremia]: isolation of virus or detection of viral protein / nucleic acid in blood samples. Including: 1CMV-DNA blood: viral DNA;2CMV antigenemia was detected in blood samples; viral DNA;2CMV antigen was detected in peripheral blood leukocytes.
  [CMV disease]: CMV infection with clinical symptoms and signs. Including: 1CMV syndrome: non-specific symptoms such as fever, fatigue, myelosuppression, elevated transaminase on the basis of CMV syndrome, and excluding fever caused by other causes and no CMV terminal organ disease; 2CMV terminal organ disease: CMV invades tissues and organs and leads to corresponding symptoms and signs (such as CMV pneumonia, CMV gastroenteritis).

SECONDARY OUTCOMES:
+30-day CMV viremia, CMV disease; +30-day overall survival, non-relapse mortality; +30-day relapse rate; +30-day aGVHD incidence. | within 30 days after allogeneic hematopoietic stem cell transplantation
  +30-day CMV viremia, CMV disease; +30-day overall survival, non-relapse mortality; +30-day relapse rate; +30-day aGVHD incidence;
+100-day overall survival, non-relapse mortality; + 100-day relapse rate; + 100-day aGVHD incidence. | within 100 days after allogeneic hematopoietic stem cell transplantation
  +100-day overall survival, non-relapse mortality; + 100-day relapse rate; + 100-day aGVHD incidence.
+180-day CMV viremia, CMV disease; +30-day overall survival, non-relapse mortality; +180-day relapse rate; +180-day aGVHD incidence. | within 180 days after allogeneic hematopoietic stem cell transplantation
  +180-day CMV viremia, CMV disease; +30-day overall survival, non-relapse mortality; +180-day relapse rate; +180-day aGVHD incidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Cao, Weijie, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes